CLINICAL TRIAL: NCT03231267
Title: Existence in the Human Digestive Flora of Phages Able to Prevent the Acquisition of Multiresistant Enterobacteria: PHAGO- BMR
Brief Title: Existence in the Human Digestive Flora of Phages Able to Prevent the Acquisition of Multiresistant Enterobacteria
Acronym: PHAGO-BMR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16011; ID RCB 2016-A01787-44 (Other: ANSM)
Record Dates: First submitted 2017-05-02; First posted 2017-07-27 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Multiresistant Enterobacteriaceae
Keywords: Multiresistant enterobacteriaceae; digestive colonization; bacteriophages; Admission in intensive care unit >72h; Presence of at least 2 consecutive stools

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "Carrier"of Ec-BLSE/EPC or Kp-BLSE/EPC: During resuscitation, evaluation of the acquisition or not of phages able to lyse Ec-BLSE / EPC or Kp-BLSE / EPC
- Non-Carrier of Ec-BLSE/EPC orKp-BLSE/EPC: During resuscitation, evaluation of the acquisition or not of phages able to lyse Ec-BLSE / EPC or Kp-BLSE / EPC

SUMMARY:
This research focuses on antibiotic resistant bacteria that may reside in the digestive tract (intestinal flora) of everyone.

When we develop an infection, the bacteria in question is, often, already present in our flora. Face to the growing phenomenon of multi-resistance, which is a public health problem, it is essential to follow the frequency of these bacteria but also to find new strategies and effective means to fight against their spread.

It has been discovered long time ago that it exists viruses able of destroying bacteria: they have been called bacteriophages .They was used before the arrival of antibiotics for the treatment of various infections (phagotherapy). Today, with the problems of resistance, phagotherapy could become a good way to fight against infections with bacteria very resistant but also a way to remove the resistant bacteria that are present in our digestive flora.

Moreover, it is known that these viruses of bacteria are present everywhere in the environment (waters, soils, human digestive tract and animal), it is important to check their presence in our digestive tract. Our objective is to study if the presence of these phages prevents resistant bacteria from set up in our digestive flora.

To answer the question, it is planned to include 460 people hospitalized in intensive care unit (resuscitation). The choice of this unit is linked to the fact that the monitoring of resistant bacteria is carried out regularly during the hospitalization. Three resuscitation services were recruited: 2 in Saint Antoine Hospital and 1 in Tenon Hospital. On stool samples collected at different times of the stay (admission and then during the stay), we will look for 2 types of bacteria and viruses capable of destroying them.

DETAILED DESCRIPTION:
Evaluate the association between the presence of phage (s) in patients not carrying E. coli or K. pneumoniae ESBL or carbapenemase (EPC) (Ec-ESBL / EPC or Kp-ESBL / EPC) and subsequent acquisition Of carrying Ec-BLSE / EPC or Kp-BLSE / EPC during their stay in intensive care.

Collection of stools of the patients included at the admission then in a successive way. On the first stool, search for multiresistant bacteria. If positive research: search for bacteriophage directed against the strain of the patient bearing. Continued screening of stools from non-carriers at baseline.

In patients defined as non-carriers at the end of the inclusions and collection, selection of 8 stools for the detection of bacteriophages directed against all BMR strains which were isolated during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admission in reanimation
* Duration of stay > 72 h.

Exclusion Criteria:

* Absence of at least 2 consecutive faeces.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients : adults admitted in intensive care for a period > 72h
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of phages capable of lysing circulating Ec-ESBL / EPC or Kp-ESBE / EPC in resuscitation units in non-carriers having acquired carriers E. coli or K. pneumoniae producing ESBL or carbapenemases . | Through study completion. An average of 1 year after the study completion.
  The classification of patients in the Carrier / Non-carrier group is based on analysis of 2 consecutive faecal samples: at least one positive sample is required to consider the patient as "carrier" of Ec-ESBL / EPC or Kp-ESBL / EPC ; It necessary to have at least 2 negative excrement to consider the patient "non-carrier. " The rate of acquisition of Ec-ESBL / EPC or Kp-ESBL / EPC will be evaluated in non-carrier patients monitored during the study.

SECONDARY OUTCOMES:
Presence or absence of phages in patients identified as carriers of Ec-ESBL / EPC or Kp-ESBL / EPC at entry to resuscitation (control population). | Through study completion. An average of 1 year after the study completion.
  Characterization of isolated phages: number and specificity (lysis capacity of one or more strains of Ec-ESBL / EPC or Kp-ESBL / EPC evaluated by the percentage of patients carrying the Ec-ESBL / EPC or Kp-ESBL / EPC ).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DECRE, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- réanimation médicale Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adhya S, Merril CR, Biswas B. Therapeutic and prophylactic applications of bacteriophage components in modern medicine. Cold Spring Harb Perspect Med. 2014 Jan 1;4(1):a012518. doi: 10.1101/cshperspect.a012518. PMID 24384811
- [Background] Balcazar JL. Bacteriophages as vehicles for antibiotic resistance genes in the environment. PLoS Pathog. 2014 Jul 31;10(7):e1004219. doi: 10.1371/journal.ppat.1004219. eCollection 2014 Jul. No abstract available. PMID 25078987